CLINICAL TRIAL: NCT01963663
Title: Comparison of Metformin and Pioglitazone Effects on Serum YKL-40 Concentrations in Patients With Newly Diagnosed Type 2 Diabetes
Brief Title: Metformin and Pioglitazone Effects on YKL-40 Concentrations in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Esteghamati, Professor Alireza Esteghamati, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 92/d/130/499
Record Dates: First submitted 2013-10-13; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: YKL-40; Chronic low grade inflammation; type 2 diabetes mellitus; metformin; pioglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator): patients receiving fixed dose metformin 1000 mg daily
  Interventions: Drug: Metformin
- Pioglitazone (Active Comparator): patients receiving fixed dose pioglitazone 30 mg daily
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Metformin — metformin 1000 mg daily in two divided doses of 500 mg tablets
  Arms: Metformin
Drug: Pioglitazone — pioglitazone 30 mg daily in two divided doses of 15 mg tablets
  Arms: Pioglitazone

SUMMARY:
Patients with type 2 diabetes are at an increased risk for developing atherosclerosis, largely due to the underlying insulin resistance and chronic low grade inflammation. Cardiovascular events could be prevented with proper interventions targeted at ameliorating the aforementioned detrimental processes. YKL-40, a novel surrogate marker of acute and chronic inflammatory states has been implicated to have a putative role in both pathways. Given the shared pathway of insulin resistance and atherosclerosis, it is conceivable that anti-diabetes medications are able to modify coronary artery disease risk via direct and indirect amelioration of YKL-40 concentrations. The present clinical trial was therefore launched to examine the comparative effects of metformin and pioglitazone, two commonly prescribed anti-diabetes medications on YKL-40 concentrations in medication-naïve, newly-diagnosed type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes patients based on American Diabetes Association criteria for diagnosis of diabetes

Exclusion Criteria:

* positive history for taking anti-diabetes medications of any class in the past
* positive current history for taking over-the-counter vitamin or anti-oxidant supplements
* presence of clinically significant chronic illnesses of the heart, lungs, or kidneys.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Serum concentration of YKL-40 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Esteghamati, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Diabetes Clinic, Vali-Asr Hospital, Tehran University of Medical Sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Esteghamati A, Azizi R, Ebadi M, Noshad S, Mousavizadeh M, Afarideh M, Nakhjavani M. The comparative effect of pioglitazone and metformin on serum osteoprotegerin, adiponectin and intercellular adhesion molecule concentrations in patients with newly diagnosed type 2 diabetes: a randomized clinical trial. Exp Clin Endocrinol Diabetes. 2015 May;123(5):289-95. doi: 10.1055/s-0034-1396864. Epub 2015 Jan 21. PMID 25607338